CLINICAL TRIAL: NCT04562064
Title: Pentacam Findings After Implantation of Intrastromal Corneal Rings in Keratoconus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: PICR
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- keratoconus group: patients with keratoconus implanted with the Myoring 360 degree, KeraRing 355 degree, KeraRing one segment, KeraRing two segments ICRS .corneal tomography scans of the two corneal surfaces were obtained preoperatively and postoperatively with a rotating Scheimpflug imaging system .pentacam data that will be included
  Interventions: Device: corneal tomography scans

INTERVENTIONS:
Device: corneal tomography scans — corneal tomography scans of the two corneal surfaces were obtained preoperatively and postoperatively with a rotating Scheimpflug imaging system

SUMMARY:
keratoconus is a progressive corneal ectatic disease characterized by paraxial stromal thinning and weakening, resulting in irregular astigmatism, corneal protrusion, and distortion of the anterior corneal surface. It is usually bilateral, although asymmetrical in most cases.

Intrastromal corneal rings are polymethylmethacrylate devices successfully used for the management of keratoconus, pellucid marginal degeneration, post-LASIK ectasia and myopia. Intrastromal corneal rings implantation is safe and reversible procedure that does not affect the central corneal area, and hence, avoids interference with visual axis. The goal of intrastromal corneal rings implantation is to improve visual acuity by regulariztion of the anterior corneal surface.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus grade I, II and III according to the mean K Amsler-Krumeich classification.
* Contact lens intolerance.
* Thinnest location is more than 400 um.
* Maximum keratometry (Kmax) between 48 and 64 D.
* Clear cornea with no Vogt's striae.

Exclusion Criteria:

* Previous corneal surgery.
* Grade IV with corneal scarring.
* Concurrent corneal disease in addition to KC.
* Autoimmune or systemic connective tissue diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with keratoconus implanted with the Myoring 360 degree, KeraRing 355 degree, KeraRing one segment, KeraRing two segments ICRS .corneal tomography scans of the two corneal surfaces were obtained preoperatively and postoperatively with a rotating Scheimpflug imaging system .pentacam data that will be included
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of changes of anterior corneal surface preoperatively compared to those values postoperativaly | 1 month
  The changes of anterior corneal surface including ﬂat (K1) and steep (K2) keratometry values, corneal astigmatism (Astig) preoperatively compared to those values postoperativaly

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No